CLINICAL TRIAL: NCT02313831
Title: Influence of Interval Aerobic Exercise Training on Cardiorespiratory and Metabolic Variables and Inflammatory Markers in Patients With Different Level of Coronary Artery Lesions
Brief Title: Optimization of Interval Exercise Based-intensity on Ventilatory Anaerobic Threshold in Coronary Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Nayara Yamada Tamburús, M.D., Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 34/2012
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Disease; Cardiovascular Risk Factors
Keywords: autonomic nervous system; ventilatory anaerobic threshold; oxygen consumption; metabolic profile; exercise training; expiratory flow limitation
MeSH Terms: conditions — Coronary Artery Disease | interventions — High-Intensity Interval Training; Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise training (Experimental): Patients of this group will be submitted to an interval training
  Interventions: Other: Interval training

INTERVENTIONS:
Other: Interval training — Patients of this group will be submitted to an interval training program
  Other Names: Cardiac rehabilitation

SUMMARY:
The purpose of this study is to investigate the effects of interval training, based-intensity on 70% at 110% of oxygen consumption and workload attained on ventilatory anaerobic threshold, on aerobic functional capacity, autonomic modulation of heart rate, metabolic profile in patients with and without coronary artery disease.

DETAILED DESCRIPTION:
Background: Exercise training has been essential component of the cardiac rehabilitation. However, it is not known if interval training based on ventilatory anaerobic threshold could be effective for improving aerobic functional capacity and metabolic profile.

Objective:To investigate the effects of interval training, based-intensity on 70% at 110% of oxygen consumption and workload attained on ventilatory anaerobic threshold, on aerobic functional capacity, autonomic modulation of heart rate, metabolic profile in patients with and without coronary artery disease.

Design: Prospective randomized controlled trial. Subjects: 68 men between 40 and 65 years old.

All subjects will be submitted:

1. - Clinical assessment: personal data, lifestyle and food, family history, current and previous history of disease.
2. - Physical examination: cardiac and lung auscultation,measurement of heart rate, blood pressure, body weight and height.
3. - Heart rate will be recorded at rest, in the supine position for 15 min, standing position for 10 min and respiratory sinus arrhythmia maneuver.
4. - Submaximal or symptom-limited cardiopulmonary exercise test on cycle ergometer will be performed to determined the ventilatory anaerobic threshold.
5. - Two cardiopulmonary exercise testing on treadmill at constant workload (moderate and high intensity). Expiratory flow limitation will be evaluated by flow-volume loops at the end of each exercise workload.
6. - Blood samples will be collected to analyze glycemic and lipid profiles.
7. - After these procedures, the subjects will be randomly assigned to one of two groups, trained group or control group.
8. - Interval training program will consist 30-40 minutes each exercise session, three times a week for 16 weeks, with a workload determined on the basis of ventilatory anaerobic threshold.
9. - At 48 hours after the last day of training, the subjects will repeat all experimental procedures as in baseline testing. Controls will be retested 16 weeks after the completion of baseline testing.
10. - All subjects will be instructed to maintain their habitual diet without a standardized caloric restriction.

Thus, it is expected that interval training will promote beneficial physiological adaptations in patients with and without coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be undergone a medical investigation for coronary artery disease, by coronary angiography, at the Hemodynamics Center of local Hospital.
* After this procedure, the CAD+ group will include 34 patients, who will have clinical evidence significant stenosis (<50% of stenosis in one or more major coronary vessels), or previous coronary artery intervention (such as percutaneous coronary intervention (PCI) and coronary artery bypass graft (CABG) surgery).
* The CAD- group will be comprised 32 patients without stenosis in coronary vessels (angiographically documented) and without history of previous myocardial infarction (MI), PCI or CABG.
* All the patients will have three or more cardiovascular risk factors such as obesity (body mass index >30 kg/m2), smoking, sedentary lifestyle according to the International Physical Activity Questionnaire (IPAQ) version 6, hypertension, diabetes mellitus (type 2 - nonusers of insulin), and dyslipidemia.

Exclusion Criteria:

* The exclusion criteria consisted of MI <6 months, PCI and CABG <3 months
* Severe cardiac arrhythmias
* Chronic obstructive pulmonary disease
* Unstable angina
* Osteomuscular disorders
* Diabetes mellitus (users of insulin)
* Renal failure
* Sequelae associated with stroke.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-01 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Intensity of interval training | 40 min
  The IT intensity levels will be prescribed based on workload (W) attained at ventilatory anaerobic threshold, i. e., at 70%, 80%, 100% and 110%

SECONDARY OUTCOMES:
Aerobic functional capacity | baseline and after interval training period (16 weeks)
  Change in oxygen consumption at ventilatory anaerobic threshold will be assessed to compare changes on oxygen uptake at baseline and after a 16 weeks of interval training.
Autonomic modulation of heart rate | baseline and after interval training period (16 weeks)
  Change in heart rate variability indices will be assessed to compare changes on cardiac parasympathetic and sympathetic modulations at baseline and after a 16 weeks of interval training.
Metabolic profile | baseline and after interval training period (16 weeks)
  Change in glycemic and lipid profiles will be assessed to compare changes in metabolic profile at baseline and after a 16 weeks of interval training.
Expiratory flow limitation | Expiratory flow limitation will be evaluated by flow-volume loops at the end of each exercise workload
  Investigate the mechanisms that limit expiratory airflow

CONTACTS AND LOCATIONS:
Overall Officials: Ester d Silva, PhD, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Nayara Yamada Tamburús, São Carlos, São Paulo, Brazil

REFERENCES:
- [Derived] Tamburus NY, Verlengia R, Kunz VC, Cesar MC, Silva E. Apolipoprotein B and angiotensin-converting enzyme polymorphisms and aerobic interval training: randomized controlled trial in coronary artery disease patients. Braz J Med Biol Res. 2018;51(8):e6944. doi: 10.1590/1414-431x20186944. Epub 2018 May 28. PMID 29846435
- [Derived] Tamburus NY, Kunz VC, Salviati MR, Castello Simoes V, Catai AM, Da Silva E. Interval training based on ventilatory anaerobic threshold improves aerobic functional capacity and metabolic profile: a randomized controlled trial in coronary artery disease patients. Eur J Phys Rehabil Med. 2016 Feb;52(1):1-11. Epub 2015 Jun 18. PMID 26086326